CLINICAL TRIAL: NCT04162509
Title: Randomized Controlled Trial on the Efficacy of a Gamified Augmented Reality Exposure-based Application in Subjects With Fear of Spiders
Brief Title: Efficacy of a Gamified Augmented Reality Exposure-based Application in Subjects With Fear of Spiders
Acronym: GARET2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-00432
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Fear of Spiders
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind study design
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly (matched by clinical relevance of fear of spiders and sex) allocated to treatment groups (experimental group, control group). The experimenter evaluating the primary outcome will be blinded (unaware of group assignment of participants, single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (Experimental): The experimental intervention in the experimental group consists of six 30-minutes AR exposures as home training (total duration in AR: 3 hours) within two weeks.
  Interventions: Other: AR app
- Control (No Intervention): The control group will not receive any active treatment (untreated comparison group).

INTERVENTIONS:
Other: AR app — Participants will be exposed to nine different AR spider scenarios with a pre-defined length of 2 minutes for each level. Each level starts with a surface scan of the environment and the placement of the AR spider model(s) by tapping on the display. Through small text pop-ups the user is instructed to perform different tasks (e.g. looking at the spider model, approaching it, holding the hand under the model). They proceed to further levels according to a predefined exposure scheme based on SUDS for fear (scale 0=no fear to 10=maximum fear) and disgust (scale 0=no disgust to 10=maximum disgust) and the assurance of the task completed (yes/no). Users will repeat each level until their SUDS are 4 or below and have completed the task. Each exposure session is limited to approx. 30 minutes (controlled by the participants) irrespective of achieved level.
  Arms: Exposure

SUMMARY:
Investigation of the efficacy of a gamified augmented reality exposure app in individual with fear of spiders.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled between subject trial. The study consists of two visits and a home training for one group. 60 participants between 18 and 40 years with clinical or subclinical fear of spiders will take part in the study.

All assessments of outcome will be conducted on one visit for each participant, including an in vivo BAT. The experimental group will participate in a home training with the app, spanning over two weeks (6x30-minutes sessions), whereas the control group will not receive any treatment (untreated comparison group).

Six weeks after the first visit all participants undergo the assessments of outcome, including a second in vivo BAT. The BAT will take place 4 weeks after completion of the home training. This design allows a direct comparison and therefore an estimation of the efficacy of the gamified AR exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fear of spiders
* BAT score before exposure between 1-8
* Physically healthy
* Fluent in German

Exclusion Criteria:

* BDI-II sumscore >=20 and/or item 9 >=1
* Concurrent psychotherapy or pharmacotherapy
* Previous exposure-based therapy for spider phobia
* Parallel participation in another study
* Chronic medication intake (except oral contraceptives)
* Medication intake before visits (less than 24h)
* Alcohol intake before visits (less than 12 h)
* Cannabis or other psychoactive substances (including benzodiazepines) intake before visits (less than 5 days)
* For women: Current pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Subjective fear (SUDS) in the in vivo BAT | 6 weeks after day one (4 weeks after completion of home training)
  During the BAT participants will be placed in front of a closed room with a spider in it and will be asked to open the door and approach a living house spider measuring about 5 cm, which will be placed in a sealed transparent plastic container on a table at the far end of the room. The participant will be requested to approach the spider and if possible, to touch the container, to remove the lid, insert a hand, and try to pick up and hold the spider for at least 20 s. Pre-defined scores ranging from 0 = refuses to enter the test room to 12 = holds the spider for at least 20 s will be given when the BAT was completed after 3 minutes or terminated by the participant. SUDS for fear and disgust will be taken during the BAT on the same score as on day one, ranging from 0 = no fear to 10 = maximum fear.

SECONDARY OUTCOMES:
Performance Behavioural Approach Test (BAT) in vivo | 6 weeks after day one (4 weeks after completion of home training)
  See primary outcome for a detailed description.
Subjective disgust (SUDS) in the in vivo BAT | 6 weeks after day one (4 weeks after completion of home training)
  See primary outcome for a detailed description.
Fear of spiders Questionnaire (FSQ) | 6 weeks after day one (4 weeks after completion of home training)
  The FSQ measures avoidance behavior as well as fear of harm and consists of 18 spider relevant situations. Participants evaluate their relationship to spiders on a 7-point Likert-type scale (0 = not at all true to 6 = absolutely true, range 0 - 108) (Szymanski and O'Donohue, 1995)
Spider Beliefs Questionnaire (SBQ) | 6 weeks after day one (4 weeks after completion of home training)
  The SBQ assesses specifically spider-related catastrophic cognitions that will be challenged within the exposure sessions and consists of 48 possible thoughts and beliefs in spider situations. Participants evaluate whether they are convinced these beliefs are true while being in a spider situation with a percentage (0 = not at all convinced to 100 = firmly convinced) (Arntz et al. 1993)
Clinical rating for specific phobia (DSM-V) | 6 weeks after day one (4 weeks after completion of home training)
  Fear of spiders will be re-assessed by the section for specific phobia (animal type: spider) of the structured diagnostic interview for mental disorders for DSM-V (DIPS, Schneider & Margraf, 2017)
Self-reported change in fear of spiders | 6 weeks after day one (4 weeks after completion of home training)
  For the self-reported change of fear of spiders participants were asked to self-rate their subjective change in fear of spiders on a single visual analogue scale in a range of 0 to 100 (0 = a lot worse, 50 = no change and 100 = a lot better).

OTHER OUTCOMES:
Self-reported change in disgust of spiders | 6 weeks after day one (4 weeks after completion of home training)
  For the self-reported change of disgust of spiders participants were asked to self-rate their subjective change in disgust of spiders on a single visual analogue scale in a range of 0 to 100 (0 = a lot worse, 50 = no change and 100 = a lot better).
AR exposure app acceptability and usability scale | 6 weeks after day one (4 weeks after completion of home training)
  The AR exposure app acceptability and usability scale consists of 11 items that assess the overall acceptability and usability (e.g. design, functionality) of the AR app for the experimental group. The items were solely composed for our study purposes. The first 9 items will be assessed through a 11-point scale, item 10 and 11 have an open answer format. Higher scores indicate higher acceptability and usability.
Credibility/Expactancy scale | On study day one
  The experimental groups therapy expectations regarding the successful treatment of their fear will be measured by an adapted credibility/expectancy for improvement scales with 5 statements. Participants rate their expectancy on a 11-point Likert-type scale (0 = not at all, 10 = absolutely, range 0 - 10) (Borkovec & Nau, 1972)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof., Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland